CLINICAL TRIAL: NCT03506672
Title: Assessing the Effectiveness of an Approach Based on the Meanings of Vocal Behaviours in Older People Living With Alzheimer's Disease in Long-term Care Facilities: DECIBELS Project
Brief Title: Assessing the Effectiveness of an Approach for Vocal Behaviors in Older People Living in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Anne Bourbonnais, Research - Chairholder, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 156273
Record Dates: First submitted 2018-04-09; First posted 2018-04-24 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Behavioral Symptoms
Keywords: Behavioral and psychological symptoms of dementia; Psychosocial interventions; Well-being; Long-term care facilities; Family and formal caregivers; Partnership
MeSH Terms: conditions — Behavioral Symptoms; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Approach based on the meanings of vocal behaviours
  Interventions: Other: Approach based on the meanings of vocal behaviours
- Control group (Active Comparator): Usual practices of formal caregivers regarding vocal behaviours
  Interventions: Other: Usual practices

INTERVENTIONS:
Other: Approach based on the meanings of vocal behaviours — Systematic problem-solving approach involving reflecting, deciding, planning and acting together (family and formal caregivers to reduce vocal behaviours and to increase everyone's well-being.
  Arms: Experimental group
Other: Usual practices — Usual practices of formal caregivers regarding vocal behaviours
  Arms: Control group

SUMMARY:
Between 13 and 60% of older people who live with Alzheimer's disease (ADRD) in long-term care facilities (LTCFs) manifest vocal behaviours (VB) that may seem inappropriate, e.g. moaning, screaming, calling out. These behaviours may indicate ill-being, disturb others, create feelings of powerlessness in family and formal caregivers, and lead to inappropriate medication. Previous efforts to reduce VB have been largely ineffective. A new approach was developed based on finding the underlying reasons for VB through a partnership between family and formal caregivers. The goals are to reduce VB, enhance older people's well-being, and increase family and formal caregivers' empowerment. The approach was tested in a pilot study of 14 triads comprising an older person living with ADRD, a family caregiver and a formal caregiver. The results were promising; overall, it is feasible to implement the approach in LTCF and it has positive effects on older people, family and formal caregivers. Now the investigators propose to assess the clinical and economic impact of the approach in 20 LTCFs with 108 triads like those in the pilot study. The approach will be implemented in 10 randomly selected "experimental" LTCFs; the other 10 (control group) will continue with their usual practices. The investigators will measure VB frequency and the well-being of the older people before, two and four months after starting the implementation. They will also measure the perceived disruptiveness of VB for family and formal caregivers, their ability to work in partnership and their empowerment relative to VB. The investigators will compare data between the control and experimental LTCFs, and calculate cost-effectiveness based on changes in VB frequency. The proposed three-year project aims to improve the well-being of all involved in LTCF by promoting a better understanding of VB and implementing a solution to optimize care. The investigators believe the findings will provide evidence to justify the wider implementation of the approach in LTCF.

DETAILED DESCRIPTION:
Aim: To assess the clinical and economic effectiveness of an approach based on the meanings of vocal behaviours (VB) in older people living with Alzheimer's disease or related disorders (ADRD) in long-term care facilities (LTCF) using a pragmatic randomized trial complemented by a qualitative component. Background: Vocal behaviours are common in LTCF; 13 to 60% of residents exhibit them. They may indicate ill-being, are associated with overmedication, are disruptive for others, and induce powerlessness in family and formal caregivers. Studies on interventions to reduce VB have shown limited clinical impacts. In previous projects, the investigators developed and pilot tested a novel approach based on the underlying meanings of VB. The systematic approach comprises family-formal caregivers' partnerships which include regular meetings (at least monthly) to identify the meanings behind VB (e.g. pain, anxiety) and to apply personalized interventions (e.g. gardening, humor). A pilot study conducted in five LTCF demonstrated the feasibility and acceptability of the recruitment and data collection methods, as well as the approach implementation using 14 triads, each made up of an older person with ADRD, a family caregiver and a formal caregiver. The approach decreased the frequency of VB, and increased the well-being of the older people with ADRD. The formal and family caregivers perceived the VB as less disruptive, and felt more empowered relative to them. However, the lack of control group precluded measuring effectiveness versus usual practices and costs. Methods: A pragmatic cluster randomized trial will be conducted to assess the effectiveness of the approach based on the results from the pilot study. A concomitant qualitative component will describe process elements that contribute to the measured effects. The investigators will randomize 20 LTCF to either an experimental (approach) or control group (usual practices), and recruit 6 triads in each LTCF for a total of 108 triads (power of 80%, significance 5%, medium effect size and 40% attrition). They will enroll 10 to 20 triads in the qualitative component. They will collect data, before, two (post-implementation) and four months (follow-up) after starting the implementation of the approach, on VB frequency (primary outcome), medication use, well-being of the older people, perceived disruptiveness of the VB, the partnership-based decision-making and the level of empowerment felt by family and formal caregivers. Additionally, they will collect data on the setting (e.g. number of beds, turnover rate), and cost (e.g. trainer, medication). Qualitative data will also be collected with individual semi-structured interviews. The investigators will analyze the effects of the approach using a mixed-model of covariance with baseline measures, and characteristics of participants and settings as covariates. They will also calculate a cost-effectiveness ratio, and do a content analysis of qualitative data. Expected outcomes: This project will provide evidence on the effectiveness of a novel and generalizable approach to increase the well-being of vulnerable older people, as well as family and formal caregivers. If effective, it may be implemented on a larger scale and adapted to other behaviours (e.g. aggressive behaviours), all of which is aligned with recommendations for research in dementia care.

ELIGIBILITY:
Inclusion Criteria:

* Older people: being 65 years old or more, having a diagnostic of Alzheimer's disease or related disorders, manifesting vocal behaviours daily and having contact with a family caregiver.
* Family caregivers: being a person that has an emotional and social relation with the older person, visiting her/him at least twice a month, speaking English or French.
* Formal caregivers: being a registered nurse (RN), licensed practical nurse (LPN), nurses' aide (NA) or another health professional involved at least three times per week in the care of the older person, speaking English or French.

Exclusion Criteria:

* Older people: having a life expectancy of less than three months
* Family caregivers: N/A
* Formal caregivers: having already participated in the trial for another older person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline frequency of vocal behaviors | 2 months
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 7-point Likert scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a high frequency; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 7

SECONDARY OUTCOMES:
Change from baseline frequency of vocal behaviors to follow-up | 4 months (follow-up)
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 7-point Likert scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a high frequency; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 7
Change from baseline in well-being | 2 months
  Quality of Life in Late-Stage Dementia (QUALID); 11 emotional states and activities on a 5-point scale; A low score indicates a better well-being; Average score Min = 11 and Max = 55
Change from baseline in well-being | 4 months (follow-up)
  Quality of Life in Late-Stage Dementia (QUALID); 11 emotional states and activities on a 5-point scale; A low score indicates a better well-being; Average score Min = 11 and Max = 55
Change from baseline in medication use | 2 months
  Medical chart
Change from baseline in medication use | 4 months (follow-up)
  Medical chart
Change from baseline in perceived disruptiveness of vocal behaviors-formal caregivers | 2 months
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 5-point disruptiveness scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a significant disruptiveness; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 6
Change from baseline in perceived disruptiveness of vocal behaviors-formal caregivers | 4 months (follow-up)
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 5-point disruptiveness scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a significant disruptiveness; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 6
Change from baseline in perceived disruptiveness of vocal behaviors-family caregivers | 2 months
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 5-point disruptiveness scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a significant disruptiveness; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 6
Change from baseline in perceived disruptiveness of vocal behaviors-family caregivers | 4 months (follow-up)
  Cohen-Mansfield Agitation Inventory (CMAI); 29 behaviours on a 5-point disruptiveness scale. Subscale "verbally agitated behaviours" of 6 items; A high score indicates a significant disruptiveness; For subscale "verbally agitated behaviours": Average score Min = 1 and Max = 6
Change from baseline in partnership-based decision-making-family caregivers' perspective | 2 months
  Family Perception of Caregiving Role (FPCR); 43 items on a 7-point Likert scale with three subscales. The sub-dimension "characteristics of the role" will be used (23 items); The lower the score, the higher is the partnership; For subscale "characteristics of the role": Average score Min = 1 and Max = 7
Change from baseline in partnership-based decision-making-family caregivers' perspective | 4 months (follow-up)
  Family Perception of Caregiving Role (FPCR); 43 items on a 7-point Likert scale with three subscales. The sub-dimension "characteristics of the role" will be used (23 items); The lower the score, the higher is the partnership; For subscale "characteristics of the role": Average score Min = 1 and Max = 7
Change from baseline in partnership-based decision-making-formal caregivers' perspective | 2 months
  Staff Perception of Caregiving Role (SPCR) questionnaire; 58 items measured on a 7-point Likert scale. Two subscales, "consequence of interactions" (32 items) and "partnership with the family" (26 items); Each one has a separate score; The lower the score, the higher is the partnership; For each subscale: Average score Min = 1 and Max = 7
Change from baseline in partnership-based decision-making-formal caregivers' perspective | 4 months (follow-up)
  Staff Perception of Caregiving Role (SPCR) questionnaire; 58 items measured on a 7-point Likert scale. Two subscales, "consequence of interactions" (32 items) and "partnership with the family" (26 items); Each one has a separate score; The lower the score, the higher is the partnership; For each subscale: Average score Min = 1 and Max = 7
Change from baseline in partnership-based decision-making-formal caregivers' attitudes | 2 months
  Attitudes about Families Checklist (AFC); 16 items measured on a 7-point Likert scale. Three subscales "quieting/disquieting" (5 items), "partner-subordinate" (4 items) and "relevant-irrelevant" (7 items); Each one has a separate score; The higher the score, the more positive is the attitude; For each subscale: Average score Min = 1 and Max = 7
Change from baseline in partnership-based decision-making-formal caregivers' attitude | 4 months (follow-up)
  Attitudes about Families Checklist (AFC); 16 items measured on a 7-point Likert scale. Three subscales "quieting/disquieting" (5 items), "partner-subordinate" (4 items) and "relevant-irrelevant" (7 items); Each one has a separate score; The higher the score, the more positive is the attitude; For each subscale: Average score Min = 1 and Max = 7
Change from baseline in empowerment-formal caregivers | 2 months
  Unique question ("When the older person manifests vocal behaviours, I feel I can do something for her/him"); 100-mm visual analogue scale ranging from Min = 0 (I feel that I cannot do anything for her/him) to Max = 100 (I feel I can always do something for her/him); The higher the score, the higher is the empowerment.
Change from baseline in empowerment-formal caregivers | 4 months (follow-up)
  Unique question ("When the older person manifests vocal behaviours, I feel I can do something for her/him"); 100-mm visual analogue scale ranging from Min = 0 (I feel that I cannot do anything for her/him) to Max = 100 (I feel I can always do something for her/him); The higher the score, the higher is the empowerment.
Change from baseline in empowerment-family caregivers | 2 months
  Unique question ("When my relative manifests vocal behaviours, I feel I can do something for her/him"); 100-mm visual analogue scale ranging from Min = 0 (I feel that I cannot do anything for her/him) to Max = 100 (I feel I can always do something for her/him); The higher the score, the higher is the empowerment.
Change from baseline in empowerment-family caregivers | 4 months (follow-up)
  Unique question ("When my relative manifests vocal behaviours, I feel I can do something for her/him"); 100-mm visual analogue scale ranging from Min = 0 (I feel that I cannot do anything for her/him) to Max = 100 (I feel I can always do something for her/him); The higher the score, the higher is the empowerment.
Cost | 2 months
  Management data

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bourbonnais, Principal Investigator — Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Locations (7):
- Canada (7):
  - CHSLD Laval et Riviera, Laval, Quebec
  - CIUSSS Nord-de-l'Île-de-Montréal, Montreal, Quebec
  - Residence Angelica, Montreal, Quebec
  - CIUSSS Ouest-de-l'Île-de-Montréal, Montreal, Quebec
  - Résidence Berthiaume-du-Tremblay, Montreal, Quebec
  - Vigi Santé, Montreal, Quebec
  - CIUSSS Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research website of principal investigator — https://www.chairepersonneagee.umontreal.ca/en/